CLINICAL TRIAL: NCT05225103
Title: Brief Suicide Intervention for Youth in Juvenile Detention Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00106321; R34MH124986 (NIH)
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Suicide Prevention
Keywords: Juvenile detention; suicidal thoughts
MeSH Terms: conditions — Suicide Prevention; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Open Trial is Single Group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SAFETY-A Implementation Sites (Experimental): New Brief Trauma-Informed Intervention (based on SAFETY-A) in addition to Enhanced Usual Care in Juvenile Detention Sites
  Interventions: Behavioral: SAFETY-Acute intervention

INTERVENTIONS:
Behavioral: SAFETY-Acute intervention — The trauma-informed brief suicide intervention based on the SAFETY-A (single crisis session in addition to follow-up caring contacts). Delivered in addition to usual care in facilities.

SUMMARY:
This is an intervention development study and therefore is not designed or powered to test hypotheses. Following initial development and refinement of intervention and protocol, an open trial will be conducted at one juvenile detention facility (n=20). Following further refinement, six juvenile detention sites will be randomized to first or second wave of intervention implementation. All youth at an implementation site in suicidal crises will receive the intervention. Data will only be collected from youth with prior assent/consent. Youth will be assessed at the time of the suicidal/self-harm crisis, and at 2 and 4 weeks after initial intervention, and at a two-month follow-up assessment. We will preliminarily examine feasibility of the intervention and associated patterns of suicidal thoughts and behavior and non-suicidal self-injury, linkage to care following release, and presumed mechanisms of change such as hopelessness, self-efficacy to remain safe, urgency to act on suicidal thoughts, and acceptance.

DETAILED DESCRIPTION:
The primary objective of this phase of the study is to develop and refine procedures for the new multi-faceted intervention for trauma-informed suicide prevention (brief cognitive-behavioral and trauma-informed strategies and safety planning for youth who are suicidal and/or self-harming, as well as training of staff in trauma-informed crisis management and de-escalation strategies) for youth in juvenile detention settings. An associated objective is to develop procedures for training staff working with youth in short-term juvenile detention settings to conduct the new intervention for reducing suicidal thoughts and behavior. A third objective is to examine the feasibility of this trauma-informed suicide prevention intervention in terms of initial participant recruitment, fidelity to the treatment model, treatment acceptability, and monitoring of adverse events in an open trial (n=20). This intervention will be iteratively refined during this open trial based on feedback from youth and staff, and experiences using the intervention in juvenile detention. We will also gather information regarding the presumed mechanisms of action and targeted outcomes for this intervention (although the small open trial will not be able to statistically examine effects).

As an intervention development study, this study is not powered to test hypotheses. Rather, the purpose of this study is to demonstrate feasibility and acceptability of the intervention and procedures, and to demonstrate viability of the proof of concept.

The study is a collaboration between Duke and Wake Forest investigators, and Juvenile Justice in the NC Department of Public Safety.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* At least 13 years of age or older and 18 years old or younger
* Without evidence from school or other records of intellectual disability
* Without evidence of active psychosis
* Not wards of the state
* Risk for suicidal behavior or non-suicidal self-harm behavior

Exclusion Criteria:

* Not English-speaking or caregivers are not English-speaking
* Wards of the state
* Younger than 13 years old or older than 18 years of age
* Evidence from school or other records or suspected intellectual disability
* Active psychosis

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2023-04-07 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Goldston, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University, Durham, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible youth were asked to assent to the study after being admitted to the facility, and parents and caregivers were then approached for consent.
Pre-assignment Details: Data were only collected from the 8 youth who were identified as being acutely suicidal and who then received the new intervention.
Units Other Than Participants: Juvenile Detention Sites
Period: Overall Study
Arm/Group | SAFETY-A Implementation Sites
Started | 8; 6 Juvenile Detention Sites
Completed | 8; 6 Juvenile Detention Sites
Not Completed | 0; 0 Juvenile Detention Sites

BASELINE CHARACTERISTICS:
Arm/Group | SAFETY-A Implementation Sites
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 0
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reported Suicide Attempts as Measured by the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: Determined by a response of "yes" to question #6 on the C-SSRS: "Have you done anything, started to do anything, or prepared to do anything to end your life?"
Time Frame: Up to 2 month follow-up assessment
Population: Data not collected on one participant.
Measure: Count of Participants; unit: Participants
Arm/Group | SAFETY-A Implementation Sites
Number analyzed (Participants) | 7
Participants | 1

2. Primary Outcome: Number of Participants Who Reported Non-Suicidal Self Injury
Description: Assessed with Questions from the Self-Injurious Thoughts and Behavior Interview.
Time Frame: Up to 2 month follow-up assessment
Population: Data not collected on one participant.
Measure: Count of Participants; unit: Participants
Arm/Group | SAFETY-A Implementation Sites
Number analyzed (Participants) | 7
Participants | 1

3. Primary Outcome: Number of Participants Who Were Linked to Mental Health Services After Release
Description: Assessed by CASA (Child and Adolescent Services Assessment) Parent Interview.
Time Frame: Up to 2 month follow-up assessment
Population: Data not collected on four participants.
Measure: Count of Participants; unit: Participants
Arm/Group | SAFETY-A Implementation Sites
Number analyzed (Participants) | 4
Participants | 3

4. Secondary Outcome: Number of Participants Reporting Urgency to Act on Suicidal Thoughts
Time Frame: Up to 2-month follow-up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | SAFETY-A Implementation Sites
Number analyzed (Participants) | 8
Participants | 1

5. Secondary Outcome: Number of Participants Reporting Hope and Reasons for Living After Leaving the Facility
Description: Adapted from items used by Cyzz et al. (2020) and Zullo et al. (2021). Number of participants who report they strongly agree that they have hope for the future and reasons for living after leaving the facility.
Time Frame: Up to 2-month follow-up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | SAFETY-A Implementation Sites
Number analyzed (Participants) | 8
Participants | 6

6. Secondary Outcome: Number of Participants Who Report Acceptance of Their Current Situation
Time Frame: Up to 2-month follow-up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | SAFETY-A Implementation Sites
Number analyzed (Participants) | 8
Participants | 7

7. Secondary Outcome: Number of Participants Reporting Self-Efficacy in Keeping Safe
Description: Adapted from items used by Czyz (2016, 2019). The number of participants reporting that they very much agreed that they felt confident in keeping themselves safe is reported.
Time Frame: Up to 2-month follow-up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | SAFETY-A Implementation Sites
Number analyzed (Participants) | 8
Participants | 6

8. Secondary Outcome: Number of Individuals With Emergency Mental Health Services (ED Visits and Hospitalizations)
Description: Assessed by CASA (Child and Adolescent Services Assessment) Parent Interview.
Time Frame: Up to 2-month follow-up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | SAFETY-A Implementation Sites
Number analyzed (Participants) | 8
Participants | 0

ADVERSE EVENTS:
Time Frame: up to 2 months
Arm/Group | SAFETY-A Implementation Sites
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAFETY-A Implementation Sites (N=8)
Suicide attempt (unverified) (Psychiatric disorders) | 1

LIMITATIONS AND CAVEATS:
As an intervention development study, this study is not powered to test hypotheses. Rather, the purpose of this study is to demonstrate feasibility and acceptability of the intervention and procedures, and to demonstrate viability of the proof of concept.

Full implementation at all but one of the facilities was challenging because of overcrowding and understaffing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-12-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT05225103/Prot_001.pdf
  • Informed Consent Form (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT05225103/ICF_000.pdf